CLINICAL TRIAL: NCT02500459
Title: A Pilot Trial of Intraparenchymally-Administered Topotecan Using Convection-Enhanced Delivery (CED) in Patients With Suspected Recurrent/Progressive WHO Grade III or IV (High Grade) Glioma Undergoing A Clinically-Indicated Surgical Resection (IND 117,240)
Brief Title: Topotecan in Glioma Undergoing A Clinically-Indicated Surgical Resection
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI Left institution
Sponsor: Michael Vogelbaum, MD, PhD (Other)
Collaborators: Infuseon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michael Vogelbaum, MD, PhD, Associate Director of the Brain Tumor and Neuro-Oncology Center, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INFT1315
Record Dates: First submitted 2015-07-15; First posted 2015-07-16 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Brain Tumor; High Grade Glioma
Keywords: Topotecan; Cleveland Multiport Catheter; Cancer
MeSH Terms: conditions — Brain Neoplasms; Glioma; Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- intraparenchymally-administered topotecan (Experimental): Patients will have topotecan administered directly into the tumor bed using convection-enhanced delivery (CED)
  Interventions: Drug: topotecan; Device: Cleveland Multiport Catheter

INTERVENTIONS:
Drug: topotecan — intraparenchymally-administered topotecan will use the Cleveland Multiport Catheter to directly infuse topotecan into the tumor site of patients with suspected recurrent/progressive high grade glioma (HGG). This drug is already FDA approved to be administered intravenously.
Device: Cleveland Multiport Catheter — The Cleveland Multiport Catheter will directly infuse topotecan into the tumor site of patients with suspected recurrent/progressive high grade glioma (HGG). Standard treatment is to adminsiter the drug intravenously.

SUMMARY:
Topotecan is an FDA-approved drug when given by intravenous infection. The purpose of this study is to determine if treatment with topotecan by an alternative method, direct delivery into the part of the brain where the tumor has spread, is safe and well tolerated. The Cleveland Multiport Catheter is a new, investigational device that will be used to deliver topotecan into tumor-infiltrated brain. A second purpose of this study is to determine whether the Cleveland Multiport Catheter can be used effectively and safely to deliver topotecan into tumor-infiltrated brain. This study will also examine how tumors responds to treatment with topotecan. This study will also look at the way topotecan is injected into tumors-infiltrated brain. A small amount of contrast dye (called gadolinium DTPA) will be added to topotecan before it is injected. Pictures will be taken of the brain with an MRI machine. This will allow the investigators to see where in the tumor-infiltrated brain the topotecan has been injected. This study will collect medical information before, during, and after treatment in order to better understand hot to make this type of procedure accessible to patients.

DETAILED DESCRIPTION:
Primary Objectives

* To investigate by magnetic resonance (MR) imaging the spatial and temporal distribution of topotecan in tumor-infiltrated brain administered by convection-enhanced delivery (CED) in patients with recurrent/progressive WHO grade III or IV (high grade) glioma (HGG) who have failed standard therapy comprising surgical biopsy and/or resection and adjuvant chemotherapy and radiotherapy, following a clinically-indicated resection of the contrast enhancing tumor mass.
* To investigate by MR imaging the influence of catheter positioning, on the spatial and temporal distribution of topotecan administered by CED in patients with recurrent/progressive HGG
* To evaluate the extent of spatial distribution of topotecan, by MR imaging, when delivered into non-enhancing tumor tissue (as defined on pre-operative conventional MRI imaging with and without intravenous gadolinium) in the intraoperative setting, the immediate peri-operative setting, and in the post-operative setting.

Secondary Objectives

* To investigate the extent to which CED-mediated delivery of topotecan
* To investigate the extent to which infusate can be distributed in the 2 cm margin around the resection cavity by administration by CED
* To assess the safety, tolerability and toxicity profile of topotecan administered by CED using different infusion rates.
* To observe evidence of activity of single-agent topotecan administered by CED to patients with recurrent/progressive HGG who have failed standard therapy comprising surgical biopsy and/or resection and adjuvant chemotherapy and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of supratentorial WHO Grade III or IV Glioma (High Grade Glioma) that has undergone surgical biopsy or resection followed by adjuvant chemoradiotherapy, that has evidence of recurrence or progression based on imaging studies and surgical resection of the enhancing tumor is clinically indicated.
* Karnofsky Performance Status 70-100;
* MRI demonstration of an enhancing mass of more than 1 cm^3 and less than 100 cm^3;
* Patient understands the procedures and agrees to comply with the study requirements by providing written informed consent; and
* Laboratory values within the following ranges:

  * Absolute neutrophil count (ANC) ≥ 1,500 / μL;
  * Platelet count ≥ 100,000 / μL;
  * Hemoglobin ≥ 10 g / dL;
  * Estimated glomerular filtration rate (eGFR) of at least 50 mL/min

Exclusion Criteria:

* Patient is mentally or legally incapacitated at the time of the study;
* Known HIV(+) or has been diagnosed with AIDS;
* Participation in another investigational drug study in the prior 4 weeks;
* Positive pregnancy test in a female;
* Patient, in the opinion of the investigator, is likely to be poorly compliant.
* Diffuse subependymal or CSF disease;
* Tumors involving the cerebellum
* Active infection requiring treatment;
* Unexplained febrile illness;
* Radiation or chemotherapy within 4 weeks of enrollment
* Systemic diseases associated with unacceptable anesthesia or operative risk;
* Personal or family history of bleeding diathesis and a coagulation profile that would preclude patient from undergoing a neurosurgical procedure
* Subject must take anticoagulants, or antiplatelet agents, including NSAIDs that cannot be stopped for surgery
* Inability to undergo magnetic resonance imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Summary of number of adverse events by grade - A measure of treatment safety | up to 1 year after start of treatment

SECONDARY OUTCOMES:
The number of patients with abnormal hematology lab reports | up to 1 year after start of treatment
The number of patients with abnormal clinical chemistry lab reports | up to 1 year after start of treatment
The number of patients with abnormal coagulation lab reports | up to 1 year after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Vogelbaum, MD, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States